CLINICAL TRIAL: NCT01842841
Title: A Multicenter, Open-label Extension Study of Velaglucerase Alfa Enzyme Replacement Therapy in Japanese Patients With Gaucher Disease
Brief Title: Multicenter Extension Study of Velaglucerase Alfa in Japanese Patients With Gaucher Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shire (Industry)
Collaborators: Quintiles, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGT-GCB-091
Record Dates: First submitted 2013-04-11; First posted 2013-04-30 (Estimated); Results first posted 2015-12-14 (Estimated); Last update posted 2021-06-14 (Actual); Status verified 2021-05

CONDITIONS: Gaucher Disease
MeSH Terms: conditions — Gaucher Disease | interventions — Glucosylceramidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- velaglucerase alfa (Experimental): 15 to 60 U/kg, EOW via intravenous infusion
  Interventions: Drug: velaglucerase alfa

INTERVENTIONS:
Drug: velaglucerase alfa — 15-60 U/kg, EOW
  Other Names: VPRIV

SUMMARY:
Gaucher disease is an inherited deficiency of the lysosomal enzyme glucocerebrosidase (GCB) that leads to progressive accumulation of glucocerebroside within macrophages and subsequent tissue and organ damage; typically of the liver, spleen, bone marrow, and brain. Type 1 Gaucher disease affects an estimated 30,000 persons worldwide and is the most common. Type 1 Gaucher disease does not involve the central nervous system. Patients with Type 2 Gaucher disease present with acute neurological deterioration, which leads to early death. Those with Type 3 disease typically display a more sub-acute neurological course, with later onset and slower progression.

The primary objective of this study is to evaluate the long-term safety of every other week (EOW) dosing of velaglucerase alfa in Japanese patients with Gaucher disease who completed study HGT-GCB-087 and elected to continue treatment with velaglucerase alfa.

Velaglucerase alfa has been developed and approved as an enzyme replacement therapy for Type 1 Gaucher disease.

DETAILED DESCRIPTION:
Gaucher disease is an inherited deficiency of the lysosomal enzyme glucocerebrosidase (GCB) that leads to progressive accumulation of glucocerebroside within macrophages and subsequent tissue and organ damage; typically of the liver, spleen, bone marrow, and brain.

Gaucher disease has been designated in the list of Specified Rare and Intractable Diseases by Specified Disease Treatment Research Program of Ministry of Health, Labor and Welfare (MHLW) as one of "lysosomal storage diseases" since 2001. Gaucher disease is also designated in the Medical Aid Program for Specified Categories of Chronic Pediatric Diseases.

The prevalence of mutations and the phenotype of patients with Gaucher disease in Japan differs from that in non-Japanese populations. Some patients with type 1 Gaucher disease in Japan have more severe and progressive disease compared to non-Japanese patients and the disease is characterized by an earlier onset of symptoms.

Velaglucerase alfa, a highly-purified form of the naturally occurring enzyme glucocerebrosidase, has been developed as an enzyme replacement therapy for Gaucher disease for the symptoms (anemia, thrombocytopenia, hepatomegaly, splenomegaly, and bone manifestation).

The primary objective of this study is to evaluate the long-term safety of every other week (EOW) dosing of velaglucerase alfa in Japanese patients with Gaucher disease who completed study HGT-GCB-087 and elected to continue treatment with velaglucerase alfa.

ELIGIBILITY:
Inclusion Criteria:

* The patient has completed treatment with EOW velaglucerase alfa through Week 51 of study HGT-GCB-087.
* Female patients of child bearing potential must agree to use a medically acceptable method of contraception at all times during the study.
* The patient, the patient's parent(s)or legal guardian(s) has provided written informed consent that has been approved by the Institutional Review Board/Independent Ethics Committee(IRB/IEC)
* The patient must be sufficiently cooperative to participate in this clinical study as judged by the Investigator.

Exclusion Criteria:

* The patient has received treatment with any investigational drug, other than velaglucerase alfa, or investigational device within 30 days prior to study entry; such use during the study is not permitted.
* The patient, patient's parent(s), or patient's legal guardian(s) is/are unable to understand the nature, scope, and possible consequences of the study.
* The patient has a significant comorbidity, as determined by the Investigator that might affect study data or confound the study results.
* The patient is unable to comply with the protocol as determined by the Investigator.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-03-13 (Actual); Primary Completion 2014-10-08 (Actual); Study Completion 2014-10-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (5):
- Japan (5):
  - Hamamatsu University School of Medicine, Hamamatsu, Shizuoka
  - Iwata City Hospital, Ōkubo, Shizuoka
  - The Jikei University School of Medicine, Minato-ku, Tokyo
  - Chiba Children's Hospital, Chiba
  - Osaka City University Hospital, Osaka

REFERENCES:
- [Derived] Ida H, Tanaka A, Matsubayashi T, Murayama K, Hongo T, Lee HM, Mellgard B. A multicenter, open-label extension study of velaglucerase alfa in Japanese patients with Gaucher disease: Results after a cumulative treatment period of 24months. Blood Cells Mol Dis. 2016 Jul;59:140-7. doi: 10.1016/j.bcmd.2015.10.002. Epub 2015 Oct 16. PMID 27241455

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants from study HGT-GCB-087 (NCT01614574) were enrolled in this study except one participant who was not enrolled due to personal reasons.
Groups:
- Velaglucerase Alfa (VPRIV®): Velaglucerase alfa (VPRIV®) 15 to 60 units per kilogram (U/kg), every other week (EOW) administered as an intravenous (IV) infusion over 60 minutes from Week 53 (2 weeks after the last infusion [Week 51] in Study HGT-GCB-087 [NCT01614574]) to Week 155.
Period: Overall Study
Arm/Group | Velaglucerase Alfa (VPRIV®)
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all enrolled participants who received at least 1 investigational product infusion (full or partial).
Groups:
- Velaglucerase Alfa (VPRIV®): Velaglucerase alfa (VPRIV®) 15 to 60 U/kg, EOW, administered as an IV infusion over 60 minutes from Week 53 (2 weeks after the last infusion [Week 51] in Study HGT-GCB-087 [NCT01614574]) to Week 155.
Arm/Group | Velaglucerase Alfa (VPRIV®)
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at the time of first dose in the current study (Week 53)
  years | 22.20 (11.946)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Drug-related Adverse Events (AEs), Infusion-related AEs, and Serious AEs (SAEs)
Description: An AE was any noxious, pathologic, or unintended change in anatomical, physiologic, or metabolic function as indicated by physical signs, symptoms, or laboratory changes occurring in any phase of a clinical study, whether or not considered related to investigational product. A SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged in-patient hospitalization; life threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. An infusion-related AE was defined as an AE that started either during or within 12 hours after the start of the infusion and that was judged as possibly or probably related to investigational product.
Time Frame: From the day of first infusion (Week 53) up to 30 days after last infusion (approximately 107 weeks)
Population: Safety population.
Measure: Number; unit: participants
Arm/Group | Velaglucerase Alfa (VPRIV®)
Number analyzed (Participants) | 5
participants
  Study drug-related AEs | 2
  Infusion-related AEs | 0
  Serious AEs | 2

2. Primary Outcome: Number of Participants Using Concomitant Medication
Time Frame: From the day of first infusion (Week 53) up to 30 days after last infusion (approximately 107 weeks)
Population: Safety population.
Measure: Number; unit: participants
Arm/Group | Velaglucerase Alfa (VPRIV®)
Number analyzed (Participants) | 5
participants | 5

3. Primary Outcome: Number of Participants With Abnormal and Clinically Significant Laboratory Test Results
Description: Laboratory test results were considered abnormal and clinically significant at the discretion of the investigator.
Time Frame: From Week 65 until the end of study (Week 155)
Population: Safety population.
Measure: Number; unit: participants
Arm/Group | Velaglucerase Alfa (VPRIV®)
Number analyzed (Participants) | 5
participants | 1

4. Primary Outcome: Number of Participants With Positive Anti-Velaglucerase Alfa Antibodies
Description: Serum samples were collected for all participants for determination of anti-velaglucerase alfa antibodies every 12 weeks.
Time Frame: From Week 65 until the end of study (Week 155)
Population: Safety population.
Measure: Number; unit: participants
Arm/Group | Velaglucerase Alfa (VPRIV®)
Number analyzed (Participants) | 5
participants | 0

5. Secondary Outcome: Change From Baseline in Hemoglobin Concentration at Week 101
Description: Baseline was the modified baseline hemoglobin concentration, the average of the values from screening, baseline, and Week 1 Day 1 from Study HGT-GCB-087 (NCT01614574).
Time Frame: Baseline, Week 101
Population: Safety population
Measure: Mean (Standard Deviation); unit: gram per deciliter (g/dL)
Arm/Group | Velaglucerase Alfa (VPRIV®)
Number analyzed (Participants) | 5
gram per deciliter (g/dL) | 0.22 (0.817)

6. Secondary Outcome: Change From Baseline in Platelet Count at Week 101
Description: Baseline was the modified baseline platelet count, the average of the values from screening, baseline, and Week 1 Day 1 from Study HGT-GCB-087 (NCT01614574).
Time Frame: Baseline, Week 101
Population: Safety population
Measure: Mean (Standard Deviation); unit: *10^9 platelets per liter
Arm/Group | Velaglucerase Alfa (VPRIV®)
Number analyzed (Participants) | 5
*10^9 platelets per liter | 9.8 (13.14)

7. Secondary Outcome: Change From Baseline in Liver Volume Normalized to Body Weight at Week 103
Description: Liver volume was measured using magnetic resonance imaging (MRI). Liver volume measurements were normalized to the percentage of body weight. Week 51 of Study HGT-GCB-087 (NCT01614574) was considered as baseline for this endpoint.
Time Frame: Baseline, Week 103
Population: Safety population
Measure: Mean (Standard Deviation); unit: Percentage of body weight
Arm/Group | Velaglucerase Alfa (VPRIV®)
Number analyzed (Participants) | 5
Percentage of body weight | 0.01 (0.207)

8. Secondary Outcome: Change From Baseline in Spleen Volume Normalized to Body Weight at Week 103
Description: Spleen volume was measured using MRI. Spleen volume measurements were normalized to the percentage of body weight. Week 51 of Study HGT-GCB-087 (NCT01614574) was considered as baseline for this endpoint.
Time Frame: Baseline, Week 103
Population: Safety population
Measure: Mean (Standard Deviation); unit: Percentage of body weight
Arm/Group | Velaglucerase Alfa (VPRIV®)
Number analyzed (Participants) | 5
Percentage of body weight | 0.04 (0.089)

9. Secondary Outcome: Change From Baseline in Bone Mineral Density (BMD) at Week 103: Z Score
Description: BMD was measured by dual energy x-ray absorptiometry (DXA) for lumbar spine and femurs. To ensure standardization and allow for comparisons of BMD, results were converted to standardized Z-scores (matched for age and gender). Z-scores express the BMD as the number of standard deviations (SDs) above or below the average BMD of a healthy participant of the same age and gender. Statistical analysis plan only required summarization if greater than (>) 50 percent (%) of participants had evaluable data. Week 51 of Study HGT-GCB-087 (NCT01614574) was considered as baseline for this endpoint.
Time Frame: Baseline, Week 103
Population: Data was not reported as there were lesser than (<) 50% of participants with evaluable data.
Arm/Group | Velaglucerase Alfa (VPRIV®)
Number analyzed (Participants) | 0

10. Secondary Outcome: Change From Baseline in Bone Mineral Density (BMD) at Week 103: T-Score
Description: BMD was measured by DXA for lumbar spine and femurs. To ensure standardization and allow for comparisons of BMD, results were converted to standardized T-scores; normal values were used from databases from Hologic based on standard criteria. T-scores are the number of SDs above or below the average for a young adult at peak BMD. Statistical analysis plan only required summarization if >50% of participants had evaluable data. Week 51 of Study HGT-GCB-087 (NCT01614574) was considered as baseline for this endpoint.
Time Frame: Baseline, Week 103
Population: Data was not reported as there were <50% of participants with evaluable data.
Arm/Group | Velaglucerase Alfa (VPRIV®)
Number analyzed (Participants) | 0

11. Secondary Outcome: Change From Baseline in Bone Marrow Burden (BMB) Score at Week 103
Description: BMB Score was measured using MRI, range from 0 (no abnormalities) to 8 points (severe disease) for the lumbar spine and from 0 (no abnormalities) to 8 points (severe disease) for the femurs. The total score was calculated as the sum of scores for femur and lumbar spine regions which ranged from 0-16 points. A higher BMB score signified more severe bone marrow involvement. Week 51 of Study HGT-GCB-087 (NCT01614574) was considered as baseline for this endpoint.
Time Frame: Baseline, Week 103
Population: Safety population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Velaglucerase Alfa (VPRIV®)
Number analyzed (Participants) | 5
units on a scale
  Lumbar spine scores | -1.2 (1.79)
  Femur scores | 0.0 (2.12)
  Total scores | -1.2 (2.95)

12. Secondary Outcome: Change From Baseline in Growth Velocity at Week 101 : Height Z-Score
Description: The Z-score, or Standard Deviation Score, is a measure of number of SDs above or below the average BMD of a healthy participant of the same age and gender. World Health Organization 2007 growth reference data were used for Z-score calculation. Statistical analysis plan only required summarization if >50% of participants had evaluable data. Week 51 of Study HGT-GCB-087 (NCT01614574) was considered as baseline for this endpoint.
Time Frame: Baseline, Week 101
Population: Data was not reported as there was <50% of participants had evaluable data.
Arm/Group | Velaglucerase Alfa (VPRIV®)
Number analyzed (Participants) | 0

13. Secondary Outcome: Change From Baseline in Skeletal Age at Week 103: Z-Score
Description: Skeletal age was measured via radiography (X-ray) of the left hand and wrist by the method of Greulich and Pyle. The Z-score, or Standard Deviation Score, is a measure of number of SDs above or below the average BMD of a healthy participant of the same age and gender. Statistical analysis plan only required summarization if >50% of participants had evaluable data. Week 51 of Study HGT-GCB-087 (NCT01614574) was considered as baseline for this endpoint.
Time Frame: Baseline, Week 103
Population: Data was not reported as there was <50% of participants had evaluable data.
Arm/Group | Velaglucerase Alfa (VPRIV®)
Number analyzed (Participants) | 0

14. Secondary Outcome: Change From Baseline in Plasma Chitotriosidase Levels at Week 101
Description: Plasma chitotriosidase activity levels were measured using an enzymatic assay with 4-methylumbelliferyl-deoxychitobiose as a substrate. Week 51 of Study HGT-GCB-087 (NCT01614574) was considered as baseline for this endpoint.
Time Frame: Baseline, Week 101
Population: Safety population. Number of participants analyzed signifies participants who were not deficient at baseline in chitotriosidase activity or who did not have a 24 base pair duplication in either copy of the chitotriosidase gene.
Measure: Mean (Standard Deviation); unit: nanomole/milliliter/hour (nmol/mL/h)
Arm/Group | Velaglucerase Alfa (VPRIV®)
Number analyzed (Participants) | 2
nanomole/milliliter/hour (nmol/mL/h) | -181.0 (268.70)

15. Secondary Outcome: Number of Participants With Change From Baseline in Neurological Status at Week 103
Description: Neurological status was considered normal or abnormal based on investigator's discretion. Week 51 of Study HGT-GCB-087 (NCT01614574) was considered as baseline for this endpoint.
Time Frame: Baseline, Week 103
Population: Safety population. Number of participants analyzed signifies participants evaluable for this outcome.
Measure: Number; unit: participants
Arm/Group | Velaglucerase Alfa (VPRIV®)
Number analyzed (Participants) | 3
participants | 0

16. Secondary Outcome: Change From Baseline in Chemokine [C-C Motif] Ligand 18 (CCL18) Levels at Week 101
Description: Plasma CCL18 concentrations were measured using a time-resolved fluorescence assay. Week 51 of Study HGT-GCB-087 (NCT01614574) was considered as baseline for this endpoint.
Time Frame: Baseline, Week 101
Population: Safety population
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Velaglucerase Alfa (VPRIV®)
Number analyzed (Participants) | 5
nanogram per milliliter (ng/mL) | -11.4 (50.97)

ADVERSE EVENTS:
Time Frame: From the day of first infusion (Week 53) up to 30 days after last infusion (approximately 107 weeks)
Arm/Group | Velaglucerase Alfa (VPRIV®)
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Velaglucerase Alfa (VPRIV®) (N=5)
Hypoacusis (Ear and labyrinth disorders) | 1 (2)
Retinal detachment (Eye disorders) | 1 (2)
Vitreous opacities (Eye disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Velaglucerase Alfa (VPRIV®) (N=5)
Hypoacusis (Ear and labyrinth disorders) | 1 (2)
Retinal detachment (Eye disorders) | 1 (2)
Vitreous opacities (Eye disorders) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Enteritis (Gastrointestinal disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Adenoiditis (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (2)
Hordeolum (Infections and infestations) | 2 (2)
Nasopharyngitis (Infections and infestations) | 2 (7)
Otitis media acute (Infections and infestations) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 2 (3)
Excoriation (Injury, poisoning and procedural complications) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Heat stroke (Injury, poisoning and procedural complications) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 1 (1)
Blood creatine phosphokinase increased (Investigations) | 1 (1)
C-Reactive protein increased (Investigations) | 1 (1)
Intraocular pressure increased (Investigations) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 3 (4)
Sleep disorder (Psychiatric disorders) | 1 (2)
Somatoform disorder (Psychiatric disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.